CLINICAL TRIAL: NCT02885870
Title: Combination of Multiparametric MRI and Electrophysiology for the Development of New Biomarkers in Spinal Cord Diseases
Acronym: SPINE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche sur la Moelle épinière et l'Encéphale (Other)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01164-45
Record Dates: First submitted 2016-08-22; First posted 2016-09-01 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Disease
Keywords: biomarker; spinal cord disease; resonance imaging; electrophysiology
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): Patient with :
  * Spinal muscular atrophy (n=25)
  * X-linked spinobulbar muscular atrophy (n=25)
  * Amyotrophic lateral sclerosis (n=25)
  Interventions: Procedure: Combination of multiparametric MRI and electrophysiology
- Healthy subject (Experimental): Subject without any neurologic or spine affection Subject matched for sex and age with patient arm
  Interventions: Procedure: Combination of multiparametric MRI and electrophysiology

INTERVENTIONS:
Procedure: Combination of multiparametric MRI and electrophysiology — MRI and electrophysiology will be combined in order to assess the human spinal cord, at both macro and microscopic levels. Specific biomarkers of white and grey matter degeneration will be developed and validated in pathologies that affect differentially white and grey matter: spinal muscular atrophy, X-linked spinal bulbar muscular atrophy and Amyotrophic lateral sclerosis

SUMMARY:
The spinal cord is a common site for the development of several neurodegenerative neurological disorders (spinal muscular atrophy or SMA, amyotrophic lateral sclerosis or ALS, X-linked spinal bulbar muscular atrophy or SBMA). In different proportions, these diseases involve axonal loss in large funiculi of the spinal white matter, their demyelination, and loss of ventral horn motor neurons or motoneurones of the spinal gray matter. The lack of specific biomarkers of these macro and microscopic spinal damages, makes it difficult the differential diagnosis and monitoring of these diseases.

Techniques to explore non-invasively the human central nervous system, such as magnetic resonance imaging (MRI) and electrophysiology, are potential tools to extract specific biomarkers of spinal damages. However, imaging techniques are still poorly developed at spinal level for technical (specific antennas), anatomical (size of the spinal cord, vertebrae) and physiological reasons (cardio-respiratory movements). However, recent advances in the field of spinal cord imaging allowed to extract quantitative data on neuron loss, axonal degeneration and demyelination in different spinal pathologies whether degenerative (ALS or SMA) or traumatic (SCI). Correlations were found with clinical data, and in ALS patients, the changes in MRI metrics over time paralleled the functional deterioration. The electrophysiological techniques are used since a long time, leading to a good knowledge of the neurophysiology of human spinal cord. In addition, electrophysiology indirectly provides data at a microscopic scale, providing information on the excitability of spinal neural networks and giving an estimate of the amount of functional neurons.

By combining these techniques for the investigation of human spinal cord in vivo, the goal is to extract new biomarkers using as study models, diseases of the spinal cord affecting differentially the white and the gray matter (SMA, SBMA and ALS).

At first, new methods of diffusion MRI and modelling will be performed in healthy subjects to assess the axonal density and diameter of the fibers in the white matter. The anatomical imaging T2 will measure the geometrical parameters of the spinal cord such as its surface and/or volume at a given vertebral level. Thanks to imaging, we will construct via methods of segmentation and image processing, an atlas of the spinal cord that will allow to locate spatially spinal atrophy in patients. After this phase of validation, A study of patients will be conducted using these new MRI techniques, in addition to those already developed in the laboratory. The contribution of electrophysiology will be to assess more accurately the microscopic damage. Quantitative data from imaging and electrophysiology will be correlated with clinical data in order to extract the most relevant biomarkers.

This project has thus a methodological interest by proposing the development of new methods to assess the human spinal cord, at both macro and microscopic levels. These methods are based on the development of the techniques developed at spinal level and which are already applicable to human pathologies. The original combination of imaging and electrophysiology will also enable us to further analyze the human spinal cord, both anatomically and functionally. This project has an important clinical value for the extraction of biomarkers in diseases where there is an unmet need for diagnosis, monitoring, prognosis and evaluation of new therapies.

ELIGIBILITY:
Inclusion Criteria

Spinal muscular atrophy patients :

* Slowly progressive weakness related to pure lower motor neuron involvement X-linked spinobulbar muscular atrophy patients
* Diagnosis confirmed by genetic testing (expansion of CAG trinucleotide repeats in the androgen receptor gene) Amyotrophic lateral sclerosis patients
* ALS definite or probable according to El Escorial criteria - No bulbar or breathing impairment preventing decubitus

Healthy volunteers

- Subjects without any neurologic or spine affection - Subjects matched for sex and age

Exclusion criteria

* Subjects not able to understand the investigator
* Subjects who are not affiliated to the national health insurance fund
* Contraindications to resonance imaging
* Contraindication to transcranial magnetic stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Change in MRI from baseline to follow-up visit | Baseline, 6 months (amyotrophic lateral sclerosis patients) or 18 months (Spinal muscular atrophy and X-linked spinobulbar muscular atrophy patients)
  Assessment of the human spinal cord, at both macro and microscopic levels. Specific biomarkers of white and grey matter degeneration.

CONTACTS AND LOCATIONS:
Locations (1):
- La Pitie Salpetrieres, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided